CLINICAL TRIAL: NCT03701685
Title: A Comparison of the Littler Flap With the Bipedicled Nerve Flap for Sensory Reconstruction of Digits
Brief Title: A Comparison of the Littler Flap With the Bipedicled Nerve Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSChen13307
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-08

CONDITIONS: Soft Tissue Defect of Digit; Nerve Injury
Keywords: nerve flap; sensory reconstruction; nerve repair

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nerve grafting (Other): The stumps of digital nerve are connected with nerve graft
  Interventions: Procedure: nerve flap

INTERVENTIONS:
Procedure: nerve flap — sensory reconstruction via a nerve graft included in the flap

SUMMARY:
A retrospective study is conducted with 59 patients who has a combination of soft tissue and digital nerve defects following trauma treated using the Littler flap or bipedicle nerve flap.Patients are divided into two groups. The group reconstructed with the Litter flap includes 26 patients and the group reconstructed with the bipedicle nerve flap includes 33 patients.Discriminatory sensation, pain and cold intolerance of the reconstructed finger, and patient satisfaction were evaluated.

DETAILED DESCRIPTION:
At final follow-up, we measured the sensation of the pulp of the reconstructed finger and the flap using the static two-point discrimination (2PD) test and Semmes-Weinstein monofilament (SWM) examination. The test points were at the centers of the radial and ulnar portions of the finger pulp and the flap. Cold intolerance of the injured and donor fingers was assessed using the self-administered Cold Intolerance Severity Score questionnaire. The maximum score was 100; scores were grouped as mild (0 to 25), moderate (26 to 50), severe (51 to 75), and extremely severe (76 to 100). Pain was given subjectively by the patient using a grading system that included grade 1, none; grade 2, mild, no interference with daily activities; grade 3, moderate, patient works but has some limitation in use of the hand because of pain; and grade 4, severe, cannot work or use hand. The Tinel sign on the donor and recipient sites was graded as follows: grade 1, none; grade 2, mild, slight tingle; grade 3, moderate, very uncomfortable; and grade 4, severe, patient unable to use hand because of any stimulation of the neuroma. Finally, patients reported their satisfaction with functional recovery of the injured finger according to the Michigan Hand Outcomes Questionnaire that was based on a 5-point response scale. All tests were performed by an independent senior hand surgeon.

ELIGIBILITY:
Inclusion Criteria:

* the defect in a region where sensory return is considered important
* soft tissue defect with exposed bone or tendon in only one digit
* associated single or double digital nerve defects with 1 to 4 cm in length7
* a soft tissue defect greater than 1.5 cm and less than 4 cm in length
* necessity to preserve digit length
* a patient between 15 and 60 years of age.

Exclusion Criteria:

* injury to the course of donor arterial pedicle or donor nerve
* nerve defect less than 1 cm or larger than 4 cm
* a soft tissue defect≤1.5 cm or ≥4 cm in length
* multiple-digit soft tissue defects
* extremely contaminated wounds
* the defect in a region the flap is unable to reach, such as thumb fingertip

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Static 2PD test | 18 months to 24 months after surgery
  We use a Disk-Criminator to test two nearby points when touching the flap. It is often

REFERENCES:
- [Result] Chen C, Tang P, Zhang L. Use of a bipedicled nerve flap taken from the dorsum of the digit for reconstruction of neurocutaneous defect in the adjacent finger. J Plast Reconstr Aesthet Surg. 2013 Oct;66(10):1322-9. doi: 10.1016/j.bjps.2013.06.001. Epub 2013 Jul 2. PMID 23829956